CLINICAL TRIAL: NCT02115386
Title: Open-label Multicenter Trial to Evaluate the Improvement of Chronic Low-grade Adverse Events Experienced by Patients With Ph+ Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) With Optimal Response to Imatinib When Switched From Imatinib to Nilotinib Treatment
Brief Title: Trial to Evaluate the Improvement of Chronic Low-grade AEs in Patients With Ph+ CML With Optimal Response to Imatinib When Switched to Nilotinib
Acronym: MACS1532
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated by Novartis
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ARU02
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Philadelphia Positive (Ph+) Chronic Myeloid Leukemia
Keywords: Ph+ CML, chronic myeloid leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nilotinib (Experimental): Dosage was 300 mg BID daily taken orally without food.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — supplied in 150 mg capsules to be taken orally

SUMMARY:
Primary Objective for this study is to evaluate changes in chronic low grade non-hematological adverse events experienced by patients who have been treated with at least 6 months of imatinib and who have not responded to supportive measures, when they are switched to nilotinib (CTCAE grading system).

DETAILED DESCRIPTION:
Study was terminated by Novartis

ELIGIBILITY:
Inclusion criteria:

Male or female patients ≥ 18 years of age 2. ECOG ≤ 2 3. Diagnosis of CML-CP < 15% blasts in peripheral blood and bone marrow

* < 30% blasts plus promyelocytes in peripheral blood and bone marrow
* < 20% basophiles in the peripheral blood
* ≥ 100 x 109 /L platelets
* No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly. 4. Minimal treatment duration before inclusion is 6 months. 5. Optimal response to imatinib at the time of inclusion according to LeukemiaNet 2009 criteria defined as:
* Patients treated with imatinib for ≥6 and <12 months must be in MCR Patients treated with imatinib for ≥12 and <18 months must be in CCR
* Patients treated with imatinib for ≥18 months must be in MMR (MMR response defined either as 3 log reduction of bcr-abl/abl ratio or as 0,1% by IS). 6. Initial treatment with 400mg imatinib with current treatment with imatinib 400 or 300 mg QD 7. Imatinib dose interruptions are allowed prior to inclusion but should not exceed 28 consecutive days 8. Persistent Grade 1- 2 non-hematological adverse events for at least 2 months despite best supportive care. Toxicity was to be evaluated by treating physician using CTCAE criteria. 9. In case of several types of non-hematological AEs no one can exceed grade 2 and at least one should last at least 2 months. 10. Adequate end organ function defined by:
* Total bilirubin < 1.5 x ULN
* AST and ALT < 2.5 x ULN
* Creatinine < 1.5 x ULN
* Serum amylase and lipase ≤ 1.5x ULN
* Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related 11. Serum potassium, magnesium, phosphorus and calcium values within normal range or corrected to within normal limits with supplements prior to first dose of study medication. 12. Patients must have an imatinib washout period of at least 3 days and not to exceed 7 days prior to the first dose of nilotinib. 13. Ability to provide written informed consent prior to any study related screening procedures being done

Exclusion criteria:

1. Patients who have experienced any Grade 3 or higher non-hematologic toxicity 30 days prior to screening
2. Loss of response (hematologic, cytogenetic, molecular) any time prior to inclusion
3. Prior accelerated phase or blast phase CML
4. Previously documented T315I mutation
5. Chromosomal abnormalities (trisomy 8) and/or clonal evolution other than Ph+.
6. Previous treatment with imatinib >400 mg any time prior to inclusion.
7. Previous treatment with any other tyrosine kinase inhibitors except for only imatinib

Impaired cardiac function including any of the following:

* LVEF < 45% as determined by echocardiogram reading or MUGA
* Complete left bundle branch block
* Long QT syndrome or a known family history of long QT syndrome
* History or presence of clinically significant ventricular or atrial tachyarrhythmias
* Clinically significant resting bradycardia (< 50 beats per minute)
* QTcF > 450 msec on baseline ECG. If QTcF > 450 and electrolytes are not within normal ranges, electrolytes were to be corrected and then the patient re-screened for QTcF
* Myocardial infarction within 1 year of starting study drug
* Other clinically significant heart disease (e.g., unstable angina, congestive heart failure, or uncontrolled hypertension) 9. Patients receiving therapy with inhibitors of CYP3A4 or medications that prolong the QT interval and cannot be either discontinued or switched to a different medication prior to starting study drug. 10. Treatment with strong CYP3A4 inducers (e.g. phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, St. John's Wort), that cannot be discontinued or switched to a different medication prior to starting study drug. 11. Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug. 12. History of acute pancreatitis within 1 year of study entry. 13. Known cytopathologically confirmed CNS infiltration (in absence of suspicion of CNS involvement, lumbar puncture not required). 14. Any other malignancy that is clinically significant or requires active intervention.

  15. Severe or uncontrolled medical conditions (i.e., uncontrolled diabetes, active or uncontrolled infection). 16. Acute or chronic liver or severe renal disease considered unrelated to cancer.

  17. History of significant congenital or acquired bleeding disorder unrelated to cancer.

  18. Previous radiotherapy to ≥ 25% of the bone marrow. 19. Major surgery within 4 weeks prior to Day 1 of study or patients who have not recovered from prior surgery. 20. Treatment with other investigational agents within 30 days of Day 1. 21. History of non-compliance to medical regimens or inability to grant consent 22. Women who are pregnant, breast feeding, or of childbearing potential without a negative urinary test at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nilotinib
Started | 7
Completed | 0
Not Completed | 7
Not completed — Protocol Violation | 1
Not completed — Administrative - trial was terminated | 6

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement of Grades of Persistent Non-hematological Adverse Event (AE) for Grade 1 and 2 at 6 Months
Description: Improvement was defined as decreasing of grade of non-hematological toxicity from 2 to <2 or from 1 to <1. In case of multiple low-grade non-hematological toxicities improvement was defined as an improvement of at least one non-hematological AE and no worsening of any other persistent non-hematological AEs.
Time Frame: at 6 month after switching from imatinib to nilotinib
Measure: Number; unit: participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 7
participants | 0

2. Secondary Outcome: Number of Participants With Improvement of Grades of Persistent Non-hematological Adverse Event (AE) for Grade 1 and 2 at 3 Months
Description: as for outcome 1
Time Frame: at 3 month after switching from imatinib to nilotinib
Measure: Number; unit: participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 7
participants | 0

3. Secondary Outcome: Number of Participants With Complete Cytogenetic Response (CCyR)
Description: Cytogenetic response will be assessed as the percentage of Ph+ metaphases in the bone marrow and is defined as the following: Complete (CCyR) - 0% Ph+ metaphases.
Time Frame: at months 6,12 and 24 after switching from imatinib to nilotinib
Measure: Number; unit: participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 6
participants | 0

4. Secondary Outcome: Number of Participants With a Major Molecular Response
Description: MMR was defined as a ≥ 3.0 log reduction in BCR-ABL transcripts compared to the standardized baseline or ≤ 0.1 % BCR-ABL/ABL % by international scale as measured by RQ-PCR, confirmed by duplicate analysis of the same sample. Molecular response was described for all time points except screening where response was estimated.
Time Frame: Months 1, 3, 6, early termination
Measure: Number; unit: participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 6
participants
  Month 1 | 5
  Month 3 | 6
  Month 6 | 6
  Early termination | 5

5. Secondary Outcome: Time to and Duration of CCyR and MMR After Switch From Imatinib to Nilotinib at 24 Months
Description: to evaluate time to achievement and duration of CCyR and MMR after switching from imatinib to nilotinib
Time Frame: at 24 Months
Population: No data collected for this Outcome Measure, as no participants reached month 24
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to First Improvement of Persistant Chronic Low-grade Non-hematologic AEs at 24 Months After Switch From Imatinib to Nilotinib
Description: Evaluate time to first improvement of low-grade non-hematologic adverse events, experienced by patients treated with imatinib and persistent despite of best supportive measures after switching to nilotinib therapy. Optimal improvement is defined as AE grade decreasing to 0.
Time Frame: first improvement of AEs after switch to 24 Months
Population: No data collected for this assessment, as no participants reached month 24
Arm/Group | Nilotinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Lisiting by Participant of EORTC-QLQ-C30 for Quality of Life
Description: EORTC-QLQ-C30 was administered to evaluate quality of life changes after switching to nilotinib. Scores ranged from 1 (very poor) to 6 (excellent)
Time Frame: Screening, months 1, 3, 6, after switch to nilotinib
Measure: Number; unit: score
Arm/Group | Nilotinib
Number analyzed (Participants) | 7
score
  Patient A Screening | 3
  Patient A Month 1 | 3
  Patient A Month 3 | 3
  Patient A Month 6 | 3
  Patient A early termination | 3
  Patient B screening | 5
  Patient B Month 1 | 5
  Patient B Month 3 | 5
  Patient B Month 6 | 5
  Patient B early termination | 5
  Patient C screening | 4
  Patient C Month 1 | 4
  Patient C Month 3 | 5
  Patient C Month 6 | 5
  Patient C early termination | 5
  Patient D screening | 3
  Patient D Month 1 | 3
  Patient D Month 3 | 3
  Patient D Month 6 | 3
  Patient D early termination | 4
  Patient E screening | 5
  Patient E early termination | 4
  Patient F screening | 4
  Patient F Month 1 | 5
  Patient F Month 3 | 5
  Patient F Month 6 | 5
  Patient F early termination | 5
  Patient G screening | 5
  Patient G Month 1 | 4
  Patient G Month 3 | 5
  Patient G Month 6 | 5
  Patient G early termination | 5

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 9 months
Groups:
- Nilotinib: Nilotinib
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=7)
HYPOACUSIS (Ear and labyrinth disorders) | 1
TINNITUS (Ear and labyrinth disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DRY MOUTH (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1
PHARYNGITIS (Infections and infestations) | 1
BILIRUBIN CONJUGATED INCREASED (Investigations) | 1
BLOOD CHOLESTEROL INCREASED (Investigations) | 1
LIPASE INCREASED (Investigations) | 2
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3
HEADACHE (Nervous system disorders) | 1
PAROSMIA (Nervous system disorders) | 1
NERVOUSNESS (Psychiatric disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.